CLINICAL TRIAL: NCT04858087
Title: Epidemiology of Malaria in Malawi: Human Hosts and Parasites in Three Districts Part 2: Cross-sectional Surveillance (School-based Cohorts)
Brief Title: Malawi International Center of Excellence in Malaria Research School-based Cohort
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Kamuzu University of Health Sciences (Other); Michigan State University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Miriam Laufer, Professor, University of Maryland, Baltimore
Other Study IDs: HP-00052129; U19AI089683 (NIH)
Record Dates: First submitted 2021-04-14; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Malaria; Malaria,Falciparum; Anemia
Keywords: cohort; screen and treat; artemether-lumefantrine
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Anemia | interventions — Mass Screening; Therapeutics; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All students: All participating students were screened for Pf infection using malaria rapid diagnostic tests (mRDTs) and treated if positive. All were followed 1, 2, and 6 weeks after screening-and-treatment.
  Interventions: Other: Screening and treatment

INTERVENTIONS:
Other: Screening and treatment — Students were screened by mRDTs and treated with artemether-lumefantrine if positive
  Other Names: mRDTs: Paracheck Orchid Biomedical Systems or SD Bioline, Standard Diagnostics Inc.; treatment with artemether-lumefantrine

SUMMARY:
A school-based, prospective, cohort study was conducted to evaluate the epidemiology of P. falciparum (Pf) infections in school-age children and determine the impact of the screen-and-treat approach on Pf infection and anemia prevalence among students in two different transmission settings. Investigators aimed to evaluate how frequently malaria rapid diagnostic tests (mRDTs) fail to detect low-parasite-density infections as well as whether low-density infections contribute to the burden and health consequences of Pf infection in school-age children and whether they contain gametocytes, the parasite stage required for transmission from humans to mosquitos.

DETAILED DESCRIPTION:
Students were enrolled in four schools in southern Malawi in the rainy (March-May) and dry season (Sept-Nov) of 2015. 15 students per grade-level (grades 1-8), were invited to participate. Following enrollment, students were evaluated at baseline for screening-and-treatment, and followed-up 1, 2 and 6 weeks later. At each follow-up visit, a blood sample was obtained for microscopy and molecular detection of parasites and students were interviewed about bed net use the night prior, current or recent illness, and use of antimalarial treatment. At the final visit, a mRDT and hemoglobin test were repeated, and parents were interviewed and portable medical records ("health passports") were reviewed to identify intercurrent fever or malaria treatment.

ELIGIBILITY:
Inclusion Criteria:

* Randomly selected student at a participating school

Exclusion Criteria:

* Parent or guardian not available for consent
* Age <5 or >= 16 years
* Known allergy or adverse reaction to lumefantrine-artemether
* Child will not attend this school during the time of the survey
* For the dry season survey (Sept-Oct 2015), participants in the rainy season survey (April-May 2015)

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 15 students per grade (1 through 8) were randomly sampled in four primary schools
Sampling Method: Non-Probability Sample
Enrollment: 786 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2015-11-13 (Actual); Study Completion 2015-11-13 (Actual)

PRIMARY OUTCOMES:
P. falciparum infection | 6 weeks after screening
  Any stage Pf infection detected by quantitative polymerase chain reaction (PCR)
P. falciparum gametocyte presence | 6 weeks after screening
  Pfs25 quantitative reverse transcriptase PCR
P. falciparum gametocyte density | 6 weeks after screening
  Pfs25 quantitative reverse transcriptase PCR

SECONDARY OUTCOMES:
Microscopic P. falciparum infection | 6 weeks after screening
  Pf infection detected by microscopy
Anemia | 6 weeks after screening
  Hb measured by Hemocue and categorized using WHO age and gender specific values

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Laufer, MD, Principal Investigator — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: Yes
data will be available via a publicly available database, such as ClinEpiDB
Supporting Information: Study Protocol
Time Frame: After results publication
Access Criteria: Public access with registration to allow tracking

REFERENCES:
- [Result] Cohee LM, Valim C, Coalson JE, Nyambalo A, Chilombe M, Ngwira A, Bauleni A, Seydel KB, Wilson ML, Taylor TE, Mathanga DP, Laufer MK. School-based screening and treatment may reduce P. falciparum transmission. Sci Rep. 2021 Mar 25;11(1):6905. doi: 10.1038/s41598-021-86450-5. PMID 33767384
- [Derived] Cohee LM, Peterson I, Buchwald AG, Coalson JE, Valim C, Chilombe M, Ngwira A, Bauleni A, Schaffer-DeRoo S, Seydel KB, Wilson ML, Taylor TE, Mathanga DP, Laufer MK. School-Based Malaria Screening and Treatment Reduces Plasmodium falciparum Infection and Anemia Prevalence in Two Transmission Settings in Malawi. J Infect Dis. 2022 Aug 12;226(1):138-146. doi: 10.1093/infdis/jiac097. PMID 35290461